CLINICAL TRIAL: NCT01361217
Title: The Effects of Multiple Dose Fluoxetine and Metabolites on CYP1A2, CYP2C19, CYP2D6 and CYP3A4 Activity
Acronym: FLUOXETINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Nina Isoherranen, Professor, PHARM: Department of Pharmaceutics, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 39288; P01GM032165 (NIH)
Record Dates: First submitted 2011-05-16; First posted 2011-05-26 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Drug-Drug Interaction; Healthy Volunteers
Keywords: Fluoxetine; CYP3A4; CYP2D6; CYP2C19; Drug-Drug Interaction; Multi-CYP Inhibition
MeSH Terms: interventions — Fluoxetine; Lovastatin; Omeprazole; Caffeine; Midazolam; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoxetine DDI (Experimental): Only arm in the study. Successive Control (Study Days 1 and 3) and fluoxetine multiple-dose treatment (Study Days 16 and 18) Sessions.
  Interventions: Drug: Fluoxetine, Lovastatin, Omeprazole, caffeine, midazolam, dextromethorphan

INTERVENTIONS:
Drug: Fluoxetine, Lovastatin, Omeprazole, caffeine, midazolam, dextromethorphan — 1x20mg oral fluoxetine capsules by mouth daily on Study Day 5, then 3x20mg fluoxetine capsules by mouth daily on Study Days 6 through 18.
  On study day 1 and study day 18, 100mg caffeine, 2mg midazolam, 30mg dextromethorphan and 20mg omeprazole (enteric coated formulation) orally with 250mL of water.
  On study day 3 and study day 20 20mg of lovastatin with 250mL of water.
  Other Names: Prozac

SUMMARY:
Inhibitory drug-drug interactions (DDIs) are a considerable concern as inhibition of drug's clearance can lead to increased plasma concentrations and subsequent adverse events and toxicities. Fluoxetine (Prozac®) is a widely prescribed antidepressant, but is also a potent inhibitor of cytochrome P450 (CYP) enzymes. Fluoxetine was chosen as the model inhibitor for this study because it is a clinically important inhibitor of multiple CYP enzymes with varying potencies for each isoform. From in vitro data, fluoxetine is predicted to be a moderate inhibitor of CYP2D6, but a strong inhibitor of CYP2C19 and CYP3A4. However, in vivo fluoxetine causes a potent interaction with CYP2D6 and a weak-to-no interaction with CYP3A4. The magnitude of the in vivo interaction of fluoxetine with CYP2C19 is not known. This in vitro-to-in vivo discrepancy is of concern for two reasons: 1) In clinical drug development, in vivo drug-drug interactions are tested only when in vitro experiments predict a risk for in vivo DDIs and 2) Because in vivo DDI's are tested using a rank order approach of going from the most potent in vitro interaction to the least potent until no interaction in vivo is observed. In this study the interaction between fluoxetine and CYP3A4, CYP2C19 and CYP2D6 will be quantified simultaneously and the quantitative in vitro-to-in vivo predictions tested. Fluoxetine will be orally administered daily for 14 days and CYP1A2, CYP3A4, CYP2C19 and CYP2D6 activity will be tested in the end of fluoxetine dosing using a cocktail of CYP probes including caffeine, midazolam, omeprazole and dextromethorphan. Lovastatin will be administered on a separate day and used as a second CYP3A4 probe to test whether CYP3A4 inhibition by fluoxetine depends on the contribution of intestinal CYP3A4 to the probe clearance. Plasma and urine samples will be collected for 12 and 24 hrs, respectively, during the control sessions (before fluoxetine administration) and for 24 hrs during the treatment sessions (fluoxetine multiple dose). The concentrations of each of the probe drugs and their metabolites (when applicable) as well as fluoxetine and its metabolites will be measured in the collected samples and pharmacokinetic analysis will be performed. The primary outcome measures for CYP inhibition will be the increase in the area under plasma concentrations time curve (AUC) of each of the probes.The null hypothesis of this study is that the area under plasma concentrations time curves (AUCs) of caffeine, dextromethorphan, omeprazole, midazolam or lovastatin are the same between the control session and the fluoxetine session. Because lovastatin has the greatest variability in its baseline pharmacokinetics the study was powered based on the specific null hypothesis for lovastatin. The alternative hypothesis is that fluoxetine decreases the clearance of the probe drugs resulting in a significant increase in the AUCs between the control and study sessions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-50 years old.
* Subjects must be currently in good health with normal gastrointestinal and heart function (as determined by medical history)
* Laboratory values indicating normal liver (Serum Albumin 3.9 - 5.0 g/dL, Total Bilirubin < 1.4mg/dL, Alanine Transaminase 9 - 60 IU/L and Aspartate Transaminase 10 - 40 IU/L) and kidney (Serum Creatinine < 1.5 mg/dL and Blood Urea Nitrogen 7 - 20 mg/dL) function as well as normal blood glucose values (Fasting Blood Glucose < 100 mg/dL).
* Subjects must have no known allergies to fluoxetine or other selective serotonin reuptake inhibitors (SSRIs), monoamine oxidase inhibitors (MAOIs), benzodiazepine drugs, caffeine, omeprazole, dextromethorphan, lovastatin or any chemically related drug.
* Women of childbearing age must be willing to use measures to avoid conception during the study period and willing to have a pregnancy test on Study Days 1 and 16.
* Subjects must agree not to take any known substrates, inhibitors, inducers or activators of cytochrome P450 (CYP) CYP1A2, CYP3A4, CYP2C19 and CYP2D6 for two weeks before the start of each study through three weeks after the last day of study. This list includes but is not restricted to antidepressant and antipsychotic agents, azole antifungal agents, macrolide antibiotics, anti-epileptic medications, antihypertensive agents and cholesterol lowering agents. They must also be willing to avoid ingesting grapefruit, grapefruit juice or other grapefruit containing products, and any herbal-based nutrient supplement or medication for the same period of time. Use of oral contraceptives will be permitted.
* Subjects must be willing to avoid caffeine-containing foods, beverages, or dietary supplements for 24 hrs prior to and throughout each study session and avoid alcohol for 48 hrs prior to and throughout each study session.
* Subjects must be willing to avoid heavy exercise during the study

Exclusion Criteria:

* Current cigarette smoker
* History of liver, kidney, gastrointestinal or heart disease
* Lab test results indicative of abnormal liver or kidney function, or diabetes (see above inclusion criteria).
* Allergy to any monoamine oxidase inhibitors (MAOIs) or any other chemically related drug or to benzodiazepine drug
* Prior experience of side effects to fluoxetine or other selective serotonin reuptake inhibitors (SSRIs)
* CYP2D6 or CYP2C19 poor metabolizer genotype or CYP3A5 expressor genotype
* Recent ingestion (< 2 weeks) of any medication known to be metabolized by or alter CYP1A2, CYP3A4, CYP2C19 or CYP2D6 activity
* A positive pregnancy test or breastfeeding
* History of diabetes, peptic ulcer or inflammatory bowel disease
* Overweight; a body mass index ≥ 30 or underweight; a body mass index of ≤ 18
* Use of chronic prescription or over-the-counter medications (except oral contraceptives)
* Use of antidepressants during the last two weeks preceding the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Isoherranen, PhD., Principal Investigator — University of Washington, School of Pharmacy, Department of Pharmaceutics; Connie Davis, MD., Principal Investigator — University of Washington, Department of Medicine

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine DDI: Only arm in the study. Successive Control (Study Days 1 and 3) and fluoxetine multiple-dose treatment (Study Days 16 and 18) Sessions.
  Fluoxetine: 1x20mg oral fluoxetine capsules by mouth daily on Study Day 5, then 3x20mg fluoxetine capsules by mouth daily on Study Days 6 through 18.
Period: Overall Study
Arm/Group | Fluoxetine DDI
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fluoxetine DDI
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  caucasian | 8
  hispanic | 1
  chicano | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
weight [Mean (Standard Deviation); unit: kg] | 72 (14)

OUTCOME MEASURES:

1. Primary Outcome: Lovastatin AUC in the Presence of Fluoxetine
Description: Our primary outcome measure will be the interaction of fluoxetine with CYP3A4. A 50% increase in the AUC for lovastatin plus hydroxy-lovastatin acid (the active form of lovastatin) between treatment day 14 (study day 20) and control days (study day 2) is considered clinically significant.
Time Frame: The primary outcome will be assessed within 2 months after the last subject is enrolled or at 2 years from the start of study enrollment, which ever is sooner.
Measure: Mean (Standard Deviation); unit: nmol*hr/L
Groups:
- Lovastatin AUC After Fluoxetine Dosing: Only arm in the study. Successive Control (Study Days 1 and 3) and fluoxetine multiple-dose treatment (Study Days 16 and 18) Sessions.
  Fluoxetine: 1x20mg oral fluoxetine capsules by mouth daily on Study Day 5, then 3x20mg fluoxetine capsules by mouth daily on Study Days 6 through 18.
- Lovastatin Before Fluoxetine: control
Arm/Group | Lovastatin AUC After Fluoxetine Dosing | Lovastatin Before Fluoxetine
Number analyzed (Participants) | 10 | 10
nmol*hr/L | 170 (70) | 180 (90)
Statistical Analysis 1: Comparison: Lovastatin AUC After Fluoxetine Dosing vs Lovastatin Before Fluoxetine; Test type: Superiority or Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Lovastatin AUC After Fluoxetine Dosing; Test type: Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: AUC of Dextromethorphan, Midazolam and Omeprazole in the Presence of Fluoxetine
Description: Our secondary outcome measure will be the interaction between fluoxetine and each CYP evaluated in the cocktail. A 50% increase in the AUC of caffeine (CYP1A2), dextromethorphan (CYP2D6), omeprazole (CYP2C19) or midazolam (CYP3A4) between treatment and control days is considered clinically significant. The interaction of fluoxetine with caffeine (CYP1A2) will be considered as a negative control for the study. These AUCs will be measured on study day 1 (control day) and study day 18
Time Frame: The secondary outcome will be assessed within 2 months after the last subject is enrolled or at 2 years from the start of study enrollment, which ever is sooner.
Measure: Mean (Standard Deviation); unit: nmol*hr/L
Groups:
- Midazolam, Caffeine, Omeprazole, Caffeine AUC After Fluoxetine: Only arm in the study. Successive Control (Study Days 1 and 3) and fluoxetine multiple-dose treatment (Study Days 16 and 18) Sessions.
  Fluoxetine: 1x20mg oral fluoxetine capsules by mouth daily on Study Day 5, then 3x20mg fluoxetine capsules by mouth daily on Study Days 6 through 18.
Arm/Group | Midazolam, Caffeine, Omeprazole, Caffeine AUC After Fluoxetine
Number analyzed (Participants) | 10
nmol*hr/L
  caffeine control AUC | 43000 (22000)
  Caffeine treatment AUC | 43000 (15000)
  dextromethophan control AUC | 68 (100)
  Dextromethorphan treatment AUC | 1850 (800)
  Omeprazole control AUC | 1200 (600)
  omeprazole treatment AUC | 8500 (3600)
  midazolam control AUC | 30 (27)
  midazolam treatment AUC | 24 (17)
Statistical Analysis 1: Comparison: Midazolam, Caffeine, Omeprazole, Caffeine AUC After Fluoxetine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Fluoxetine DDI
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine DDI (N=10)
anxiety (Psychiatric disorders) | 1 (1) — One subject experienced an anxiety attack during the study. No other adverse events reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No